CLINICAL TRIAL: NCT00981435
Title: Steroids And Laser Trabeculoplasty (SALT) Trial: Effect of Anti-Inflammatory Treatment on the Efficacy of SLT
Brief Title: Steroids After Laser Trabeculoplasty for Glaucoma
Acronym: SALT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Bascom Palmer Eye Institute (Other); University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20081142
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Glaucoma
Keywords: Glaucoma; Trabeculoplasty; Selective laser trabeculoplasty; Intraocular pressure
MeSH Terms: conditions — Glaucoma | interventions — 1(beta)-D-arabinofuranosylcytosine-5'-diphosphate prednisolone; prednisolone acetate; Ketorolac; Diclofenac; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Artificial Tears (Experimental): Topical artificial tears dosed 4 times per day for 4 days in treated eye after laser trabeculoplasty.
  Interventions: Drug: Artificial Tears
- Non-steroidal anti-inflammatory (Experimental): Topical ketorolac 0.5% dosed 4 times per day for 4 days in treated eye after laser trabeculoplasty.
  Interventions: Drug: Ketorolac
- Steroid (Experimental): Topical prednisolone 1% dosed 4 times per day for 4 days in treated eye after laser trabeculoplasty.
  Interventions: Drug: Prednisolone 1%

INTERVENTIONS:
Drug: Prednisolone 1% — Prednisolone 1% to lasered eye 4 times/day for 4.5 days
  Other Names: Pred forte
  Arms: Steroid
Drug: Ketorolac — Ketorolac 0.5% to lasered eye 4 times/day for 4.5 days
  Other Names: Voltaren
  Arms: Non-steroidal anti-inflammatory
Drug: Artificial Tears — Artificial saline tears to lasered eye 4 times/day for 4.5 days
  Other Names: saline tears
  Arms: Artificial Tears

SUMMARY:
The purpose of this study is to determine whether the choice of post-operative eye drop administered after selective laser trabeculoplasty (SLT) for glaucoma affects the efficacy in lowering intraocular pressure (IOP).

DETAILED DESCRIPTION:
SLT is used to lower intraocular pressure in glaucoma, but it is not know whether the choice of eyedrops administered in the post-operative period affects SLT efficacy. Practitioners commonly use steroid drops, non-steroidal anti-inflammatory drops, or no drops at all. This is a randomized, single-center, prospective, masked clinical trial to determine whether the choice of eyedrop affects efficacy of SLT in glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of glaucoma
* clinician has determined that SLT laser is indicated
* IOP currently >18 and was ever >21 in the past (e.g. prior to treatment)

Exclusion Criteria:

* prior history of uveitis
* prior glaucoma surgery including glaucoma laser surgery
* pregnant or 3 months post-partum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2009-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey L Goldberg, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Bascom Palmer Eye Institute, Miami, Florida
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
IPD is anticipated to be shared upon publication of results.

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-steroidal Anti-inflammatory: Diclofenac 0.1%: Diclofenac sodium 0.1% to lasered eye 4 times/day for 4.5 days
Period: Overall Study
Arm/Group | Artificial Tears | Non-steroidal Anti-inflammatory | Steroid
Started | 31 | 29 | 37
Completed | 31 | 29 | 37
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Artificial Tears | Non-steroidal Anti-inflammatory | Steroid | Total
Number analyzed (Participants) | 31 | 29 | 37 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (15) | 60 (11) | 67 (14) | 65 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 23 | 56
  Male | 12 | 15 | 14 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 5 | 11 | 26
  Not Hispanic or Latino | 20 | 23 | 24 | 67
  Unknown or Not Reported | 1 | 1 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 7 | 8 | 21
  White | 25 | 21 | 29 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) Change
Description: IOP will be measured before and at 6 and 12 weeks after intervention using Goldman tonometry.
Time Frame: Baseline to Week 12
Population: Patient data was incomplete due to inadequate measurement or follow up as follows: Artificial tears (31 enrolled, 27 available at 6 weeks, 25 at 12 weeks); Non-steroidal anti-inflammatory (28 enrolled, 27 available at 6 and 12 weeks); Steroid (37 enrolled, 33 available at 6 weeks, 29 at 12 weeks).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Artificial Tears | Non-steroidal Anti-inflammatory | Steroid
Number analyzed (Participants) | 25 | 27 | 29
mmHg | -3.0 (4.3) | -6.2 (3.1) | -5.2 (2.7)

2. Secondary Outcome: Intraocular Inflammation
Description: The count of patients with inflammation defined as anterior chamber cells was measured in each study arm.
Time Frame: Up to week 12
Population: Patient data was incomplete due to inadequate measurement or follow up as follows: Artificial tears (31 enrolled, 31 available for data acquisition); Non-steroidal anti-inflammatory (29 enrolled, 26 available for data acquisition); Steroid (37 enrolled, 35 available for data acquisition).
Measure: Count of Participants; unit: Participants
Arm/Group | Artificial Tears | Non-steroidal Anti-inflammatory | Steroid
Number analyzed (Participants) | 31 | 26 | 35
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: Adverse events and serious adverse events were pre-defined and evaluated by examining physician at every study visit.
Arm/Group | Artificial Tears | Non-steroidal Anti-inflammatory | Steroid
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/37
Other Adverse Events (participants affected / at risk) | 0/31 | 0/29 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No